CLINICAL TRIAL: NCT02171117
Title: Phase III Clinical Trial of Microtransplantation to Treat Elderly Acute Myeloid Leukemia
Brief Title: Safety and Efficacy Study of Microtransplantation to Treat Elderly Acute Myeloid Leukemia
Acronym: IMCG-EAML
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Affiliated Hospital of the Chinese Academy of Military Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IMCG-EAML2014
Record Dates: First submitted 2014-06-17; First posted 2014-06-24 (Estimated); Last update posted 2016-07-13 (Estimated); Status verified 2016-07

CONDITIONS: Acute Myeloid Leukemia
Keywords: Acute Myeloid Leukemia; microtransplantation; elderly patients; HLA-mismatched; donor; Peripheral; stem cell; infusion
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CT-group (No Intervention): standard induction and consolidation chemotherapy only, without microtransplantation
- MST-group (Experimental): standard induction and consolidation chemotherapy with microtransplantation
  Interventions: Procedure: microtransplantation; Biological: HLA-mismatched donor peripheral stem cell infusion

INTERVENTIONS:
Procedure: microtransplantation — infusion of granulocyte colony stimulating factor (G-CSF) mobilized HLA-mismatched peripheral blood stem cells (GPBSC)
  Other Names: DSI
  Arms: MST-group
Biological: HLA-mismatched donor peripheral stem cell infusion
  Arms: MST-group

SUMMARY:
Patients enrolled from each center according to confirmed criteria specified in cooperative scheme are randomly assigned to standard induction and consolidation chemotherapy with microtransplantation （MST-group）or without (CT-group).Compare the remission rate and 2-year disease-free survival (DFS) and overall survival(OS) rate of the two groups.

DETAILED DESCRIPTION:
Microtransplantation, which combines chemotherapy with adoptive infusion of granulocyte colony stimulating factor (G-CSF) mobilized HLA-mismatched peripheral blood stem cells (GPBSC). Data from more than 70 elderly AML patients who received microtransplantation in Beijing showed that the remission rate and 2-year disease-free survival (DFS) reach 75-82% and 32-39% respectively, and microchimerisms (donor cells<1%) were detected without GVHD. The results have been clinically validated in several other centers in China, United States and Australia. Based on these facts, to further validate the therapeutic efficacy, we propose a phase III clinical trial in which the de novo AML patients ≥60 years old are randomly assigned to receive standard induction and consolidation chemotherapy with or without microtransplantation.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have elderly (60-85 ages) AML pathologically confirmed per WHO guidelines.
* Patients have not been treated before.
* Patients must have ECOG Performance status of 0,1,or 2. If ECOG 2.
* Patients must have a HLA mismatched donor who should be able to provide informed consent.
* All genders and races are eligible.
* ALT and AST≤3 ×ULN, TBIL≤1.5 × ULN, Cr≤2 ×ULN or CrCl≥40 mL/min
* By means of ultrasonic Heartbeat map or multiple gated acquisition (MUGA) scanning determination of LVEF in the normal range.
* Donors must be able to safely undergo leukapheresis.

Exclusion Criteria:

* received operation 4 weeks before randomization
* acute promyelocytic leukemia,Myeloid sarcoma, chronic myeloid leukemia in accelerated phase and blastic phase;
* active CNS disease, pregnancy, or other major medical or psychiatric illnesses that could compromise tolerance to this protocol
* occurred stroke or intracranial hemorrhage within 6 months before randomization.
* Require the use of warfarin or equivalent of vitamin K antagonists (such as phenprocoumon) anticoagulant.
* There is clinical significance of cardiovascular disease, such as uncontrolled or symptomatic arrhythmias, congestive heart failure or myocardial infarction within 6 months before randomization, or any heart function grade 3 (moderate) or 4 (severe ) heart disease in accordance with the functional classification method of New York Heart Association (NYHA).
* Known to have the following history: human immunodeficiency virus (HIV) or active hepatitis C virus or hepatitis B virus infection
* Any situation processed by the PI that will be damaged to the patients safety.
* Patients and / or authorized family member refuse to sign the consent.
* attend other clinical researchers in 3 months.
* Donors exclusion criteria include:active infection or malignancy, cardiovascular instability, severe anemia, severe coagulation disorder, pregnancy, inadequate venous access, inability to provide consent, or any other condition deemed unsafe by the treatment staff.

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 196 (Estimated)
Dates: Start 2014-03; Primary Completion 2018-06 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
the remission rate | 2 months
  ①bone marrow: blasts <5% (with a count of at least 200 Nucleated cells).②Hemogram: absolute neutrophil count of more than 1.0×109/L，platelets of >100×109/L. ③Clinical: Without the signs and symptoms caused by leukemia infiltration d , and independent of transfusion;

SECONDARY OUTCOMES:
Disease Free Survival | 2 years
  Measured from complete remission to the date of death or the date of last follow-up examination;
Overall Survival | 2 YEAR
  measured from the Date of beginning therapy to the date of death or the date of last follow-up examination;

OTHER OUTCOMES:
treatment-related mortality | 2 years
  Early mortality: death within 4 weeks after initiation of induction therapy
donor chimerism or microchimerism | at count recovery prior to each new cycle of therapy, at 4 weeks after the last round of consolidation, and if still positive, every 3 months after completing therapy for up to 2 years
donor versus leukemia effect | 2 years
  Analysis of donor WT1 positive CD8 T cells by flow cytometry
recipient versus leukemia effect | 2 YEAR
  Analysis of recipient WT1 positive CD8 T cells by flow cytometry

CONTACTS AND LOCATIONS:
Overall Officials: AI HUISEHNG, MD, Principal Investigator — Affiliated Hospital of Academy of Military Medical Sciences
Locations (1):
- Affiliated Hospital of Academy of Military Medical Sciences ,, Beijing, Beijing Municipality, China